CLINICAL TRIAL: NCT03274791
Title: Airway Inflammatory Profile and Clinical Presentation of COPD: A Comparison Between Never Smokers and Smokers
Brief Title: Clinical Features and Airways Inflammation in Never Smokers and Smokers With COPD
Status: Completed | Type: Observational
Sponsor: Ministry of Scientific Research, Tunisia (Other Government)
Responsible Party: Principal Investigator, Myriam Denguezli, Assistant Professor, Ministry of Scientific Research, Tunisia
Other Study IDs: COPDNS
Record Dates: First submitted 2017-08-24; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: COPD; Airway Obstruction; Inflammation
Keywords: COPD; smoking; induced sputum; clinical features
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Airway Obstruction; Inflammation; Smoking | interventions — Respiratory Function Tests; Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy subjects: Healthy non-smoking subjects were never smokers with normal spirometry and did not have a history of lung disease or chronic respiratory symptoms.
  Information about respiratory symptoms and comorbidities were collected. Healthy subjects underwent pulmonary function tests (Spirometry). Induced sputum was collected to determine total and differential inflammatory cells counts as well as inflammatory mediators (Interleukin-8 and tumor necrosis factor-alpha).
  Interventions: Diagnostic Test: Analysis of induced sputum; Diagnostic Test: Lung Function test; Diagnostic Test: Enzyme-linked Immunosorbent Assay
- COPD Never smokers: Never smokers referred to subjects who had never smoked Airflow limitation in COPD was defined as a post-bronchodilator forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) ratio <70% and FEV1 reversibility of <12% and 200 mL from baseline values after inhalation of 400 µg of Salbutamol.
  Information about respiratory symptoms and comorbidities were collected. Never smoking subjects with COPD underwent pulmonary function tests (Spirometry). Induced sputum was collected to determine total and differential inflammatory cells counts as well as inflammatory mediators (Interleukin-8 and tumor necrosis factor-alpha).
  Interventions: Diagnostic Test: Analysis of induced sputum; Diagnostic Test: Lung Function test; Diagnostic Test: Enzyme-linked Immunosorbent Assay
- COPD Smokers: Smokers were defined as persons who had smoked > 20 packs of cigarettes in a lifetime and who continue smoking every day.
  Airflow limitation in COPD was defined as a post-bronchodilator forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) ratio <70% and FEV1 reversibility of <12% and 200 mL from baseline values after inhalation of 400 µg of Salbutamol.
  Information about respiratory symptoms and comorbidities were collected. Smoking subjects with COPD underwent pulmonary function tests (Spirometry). Induced sputum was collected to determine total and differential inflammatory cells counts as well as inflammatory mediators (Interleukin-8 and tumor necrosis factor-alpha).
  Interventions: Diagnostic Test: Analysis of induced sputum; Diagnostic Test: Lung Function test; Diagnostic Test: Enzyme-linked Immunosorbent Assay

INTERVENTIONS:
Diagnostic Test: Analysis of induced sputum — Induced sputum was collected and analysed in the three arms (Healthy subjects, Never smokers with COPD and smokers with COPD) The volume of the sputum sample, was treated with an equal volume of 0.1% dithiothreitol. The samples were then vortexed and placed in a shaking water bath at 37°C for 15 min to ensure complete homogeneisation. The suspensions were centrifuged at 400× g and the sputum supernatant stored at -80°C until cytokines analysis. The cell pellet was resuspended in 0.5% bovine serum albumin in phosphate buffered saline and cytospin were made by putting 100 µL of the cell suspension in the funnels.
  Slides for differential cell counts were stained with May-Grünwald Giemsa.
Diagnostic Test: Lung Function test — All the subjects underwent pulmonary function tests (Healthy subjects, Never smokers with COPD and smokers with COPD).
  Pulmonary function parameters were measured using a portable spirometer (Easy One ndd. Medizintechnik; Zurich, Switzerland) according to the ATS criteria (American Thoracic Society). Reversibility test was performed 15 min after inhalation of 400 µg of Salbutamol (Ventolin, GlaxoSmithKline, Middlesex, UK). All spirometry data were graded for quality and only tests that met high quality scores were used for the final analysis.
  Other Names: spirometry
Diagnostic Test: Enzyme-linked Immunosorbent Assay — IL-8 and TNF-α were measured in the sputum supernatant of all the subjects (Healthy subjects, Never smokers with COPD and smokers with COPD).
  Commercially available kits were used to detect IL-8 (Human IL-8 Immuno-Biological Laboratories ELISA Kit) and TNF-α (Human TNF-alpha Sigma-Aldrich ELISA Kit) concentrations in the sputum supernatants. The absorbance was measured at 450 nm. The lower limits detection were 2 pg/mL for IL-8 and 5 pg/mL for TNF-α. The intra assay coefficients of variability were 8.7% for IL-8 and 7.7% for TNF- α.
  Other Names: ELISA

SUMMARY:
The aim of this study was to investigate the airway inflammatory profile and the clinical presentation of chronic obstructive pulmonary disease (COPD) in never smokers compared to smokers with COPD.

DETAILED DESCRIPTION:
40 COPD patients (21 smokers and 19 never smokers) and 28 healthy never smokers were included in the present study. Information about respiratory symptoms and comorbidities were collected. Subjects underwent pulmonary function tests and COPD was defined according to Global Initiative for Chronic Obstructive lung Disease spirometric criteria. Induced sputum was collected to determine total and differential inflammatory cells counts as well as inflammatory mediators (Interleukin-8 (IL-8) and tumor necrosis factor-alpha (TNF-α)). The Mann-Whitney U and the χ2 tests were used for results comparisons. Correlations between symptoms, spirometric parameters, cytokines levels, inflammatory cells and risk factors of COPD were examined with Spearman's rank correlation test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with COPD, according to GOLD criteria (smokers and never smokers). Moreover, inhaled short-acting β2-agonists were stopped at least 8h before the test and inhaled long-acting β2-agonist were stopped at least 48h before the test.
* Healthy control subjects : never smokers with normal spirometry and did not have a history of lung disease or chronic respiratory symptoms.

Exclusion Criteria:

* COPD patients were excluded from the study if they had an exacerbation, a respiratory tract infection or if they used a systemic form of corticosteroid preparation (oral or intravenous injection therapy) or antibiotics within the two months prior to the study entry. Patients with other respiratory disorder like pneumonia, pulmonary emboli, congestive heart failure, lung cancer or tuberculosis were also excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the department of physiology and functional explorations of Sousse University Hospital. 40 subjects with COPD, according to GOLD criteria (21 current smokers and 19 never smokers) and 28 healthy control subjects participated to the study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Weight measurement | 6 months
  Weight was measured in kilograms for all the participants.
Height measurement | 6 months
  Height was measured in meters for all the participants.
Forced vital capacity (FVC) | 6 months
  FVC was measured using a portable spirometer (Easy One ndd. Medizintechnik; Zurich, Switzerland) according to the American Thoracic Society criteria.
Forced expiratory volume in one second (FEV1) | 6 months
  FEV1 was measured using a portable spirometer (Easy One ndd. Medizintechnik; Zurich, Switzerland) according to the American Thoracic Society criteria.
Sputum induction and collection | 6 months
  Sputum induction was conducted by inhalation of nebulised sterile hypertonic saline solution followed by coughing and expectoration of airway secretions. For nebulisation, an ultrasound nebulizer was used for 5-20 min to provide an adequate amount of sample. The subject is asked to cough and expectorate at 5 min intervals.

SECONDARY OUTCOMES:
BMI determination | 6 months
  Weight and height values were combined to report BMI in kg/m2
Tiffeneau ratio (FEV1/FVC) | 6 months
  The calculation of FEV1/FVC allows the identification of obstructive ventilatory defect. A FEV1/FVC < 70 % where FEV1 is reduced more than FVC signifies an obstructive defect.
Sputum cell counts | 1 month
  Four hundred non-squamous cells were counted by two technicians and the mean of the two scores was expressed as percentage of the total cell count. Sputum samples containing >20% of squamous cells and/or with cell viability <70% were excluded from analysis.
Sputum supernatant analyses | 3 months
  IL-8 and TNF-α sputum supernatant concentrations were measured in the sputum supernatant of the three studied groups using ELISA test.

CONTACTS AND LOCATIONS:
Overall Officials: Zouhair Tabka, MD PhD, Study Director — Faculty of Medicine of Sousse; Amina Mrizak, MSc, Principal Investigator — Faculty of Medicine of Sousse

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results will be shared in a publication
Supporting Information: Study Protocol, CSR
Time Frame: The data will become available when the article will be accepted by the editorial board of the journal.